CLINICAL TRIAL: NCT02950987
Title: Screening With Whole Body MRI For Detection Of Primary Tumors In Children And Adults With Li-Fraumeni Syndrome (LFS) And Other Cancer Predisposition Syndromes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Allison O'Neill, MD, Instructor, Pediatric Hematology/Oncology, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 11-200
Record Dates: First submitted 2016-10-11; First posted 2016-11-01 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Li-Fraumeni Syndrome
Keywords: Li-Fraumeni Syndrome (LFS); Cancer Predisposition Syndromes; LFS
MeSH Terms: conditions — Li-Fraumeni Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Whole Body MRI (Experimental): * Magnetic resonance imaging will be performed on participants
  * Participants who are two young to tolerate the scans awake, can receive sedation/anesthesia
  Interventions: Device: Whole Body MRI

INTERVENTIONS:
Device: Whole Body MRI

SUMMARY:
This study is evaluating Whole Body MRI as a possible screening tool to diagnose cancer for people with LFS and other inherited cancer predisposition syndromes.

DETAILED DESCRIPTION:
Individuals who carry the TP53 mutation have a higher risk of developing different types of cancer over their lifetimes. This gene has been associated with Li Fraumeni syndrome in some families, but not all families that have cancer histories consistent with Li Fraumeni syndrome will have the mutation. Currently, there is no standard method of monitoring LFS carriers, family members, or others individuals with cancer predisposition syndromes to detect cancers in the early stages, when they may be more easily treated.

The main aim of the study is to test a relatively new medical technology called Whole Body Magnetic Resonance Imaging (MRI), in patients with these syndromes, to see if cancers can be detected at an early stage which may, in turn, allow for more effective treatment. The investigators have chosen Whole Body MRI scanning because this scan allows doctors to look at the entire body in one examination. By using this technology, participants are not exposed to radiation, which is of particular importance for individuals who have a higher cancer risk due to a diagnosis of LFS.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Individuals greater than or equal to 18 years of age.
* Individuals with "Li Fraumeni Syndrome" defined as one of the following:

  * Carriers of a germline p53 mutation
  * Members of families meeting classic LFS criteria by family history without an identifiable p53 mutation
  * Obligate carrier by pedigree (these individuals can be offered testing but are still eligible if they defer). The following examples describe "obligate carriers by pedigree."
* A child of a parent with known p53 mutation that is diagnosed with cancer
* An individual with a sibling and a child who are p53 positive -OR-
* Individuals with an inherited cancer predisposition syndrome as defined by one of the following:

  * Hereditary Retinoblastoma with a germline Rb mutation
  * Diagnosis of Hereditary Paraganglioma/Pheochromocytoma Syndrome with a germline SDH mutation
  * Diagnosis of Multiple Endocrine Neoplasia, Type 1 or 2, with a germline MEN mutation
  * New diagnosis of opsoclonus-myoclonus with a negative cancer work-up upon presentation of symptoms
  * Familial Neuroblastoma with a germline ALK mutation
  * Rapid-onset Obesity with Hypothalamic dysfunction, Hypoventilation and Autonomic Dysregulation (ROHHAD syndrome) or Congenital central hypoventilation syndrome (CCHS) with or without a germline PHOX 2B mutation
  * Von Hippel-Lindau with a VHL mutation
  * Women with an abnormal cell-free DNA test (i.e. a non-invasive prenatal test (NIPT) to detect chromosomal abnormalities) and no cancer diagnosis
  * Other rare cancer predisposition syndromes at the discretion of the treating physician and study physicians
* NOTE: Individuals with any of the above-listed cancer predisposition syndromes (apart from Li Fraumeni syndrome) are likewise eligible in the absence of a known mutation if they are an obligate carrier by pedigree.
* Individuals can have a prior history of cancer; these individuals must be in stable remission and at least 6 months out from the completion of surgery/radiation\ therapy/chemotherapy.
* Individual cases can be reviewed with the institutional principal investigator.
* Individuals not pregnant at enrollment. Female subjects of childbearing potential will undergo a pregnancy test prior to imaging.
* Individuals able to give informed consent or a signature from a designated health care proxy or legal guardian.

Children

* Individuals who are less than 18 years of age
* Individuals with "Li Fraumeni Syndrome" defined as one of the following:

  * Carriers of a germline p53 mutation OR
  * Members of families meeting classic LFS criteria by family history without an identifiable p53 mutation OR
  * Obligate carrier by pedigree (these individuals can be offered testing but are still eligible if they defer). The following examples describe "obligate carriers by pedigree."
* A child of a parent with known p53 mutation that is diagnosed with cancer
* An individual with a sibling and a child who are p53 positive -OR-
* Individuals with an inherited cancer predisposition syndrome as defined by one of the following:

  * Hereditary Retinoblastoma with a germline Rb mutation
  * Diagnosis of Hereditary Paraganglioma/Pheochromocytoma Syndrome with a germline SDH mutation
  * Diagnosis of Multiple Endocrine Neoplasia, Type 1 or 2, with a germline MEN mutation
  * New diagnosis of opsoclonus-myoclonus with a negative cancer work-up upon presentation of symptoms
  * Familial Neuroblastoma with a germline ALK mutation
  * Rapid-onset Obesity with Hypothalamic dysfunction, Hypoventilation and Autonomic Dysregulation (ROHHAD syndrome) or Congenital central hypoventilation syndrome (CCHS) with or without a germline PHOX 2B mutation
  * Von Hippel-Lindau with a VHL mutation
  * Other rare cancer predisposition syndrome at the discretion of the treating physician and study physicians
* NOTE: Individuals with any of the above-listed cancer predisposition syndromes (apart from Li Fraumeni syndrome) are likewise eligible in the absence of a known mutation if they are an obligate carrier by pedigree.
* Individuals can have a prior history of cancer; these individuals must be in stable remission and at least 6 months out from the completion of surgery/radiation therapy/chemotherapy. Individual cases can be reviewed with the institutional principal investigator.
* Individuals not pregnant at enrollment. Female subjects of childbearing potential will undergo a pregnancy test prior to imaging.
* Signed document of informed consent completed by the parent or legal guardian
* Signed document of assent obtained if child ≥10 years of age

Exclusion Criteria:

Adults and Children

* Active cancer or metastatic disease, except in the case of Stage 0 Chronic Lymphocytic Leukemia or nonmelanoma skin cancer.
* Patients with a contraindication to sedation or general anesthesia
* Patients with a metal heart valve, surgical clips, a pacemaker or any other indwelling metal device that might interfere with MRI
* Females who are pregnant or nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Return of pediatric and adult patients with Li Fraumeni Syndrome year-after-year for 4 annual scans. | 4 years
  Successful return of patients for four annual scans will be recorded.

SECONDARY OUTCOMES:
Return of pediatric and adult patients with other cancer predisposition syndromes year-after-year for 4 annual scans. | 4 years
  Successful return of patients for four annual scans will be recorded.
Detection of prevalent and incident cancers on WB-MRI in pediatric and adult patients with Li Fraumeni and other inherited cancer predisposition syndromes. | 3 years
  Tabulation of all follow-up imaging studies, biopsies, and cancer diagnoses will be pursued.
Detection of prevalent and incident cancers on additional screening studies in pediatric and adult patients with Li Fraumeni and other inherited cancer predisposition syndromes. | 3 years
  Tabulation of all follow-up imaging studies, biopsies, and cancer diagnoses will be pursued.

CONTACTS AND LOCATIONS:
Overall Officials: Allison O'Neill, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No